CLINICAL TRIAL: NCT01779206
Title: Adjuvant Dynamic Marker-Adjusted Personalized Therapy Trial Optimizing Risk Assessment and Therapy Response Prediction in Early Breast Cancer
Brief Title: ADAPT - Adjuvant Dynamic Marker-Adjusted Personalized Therapy Trial Optimizing Risk Assessment and Therapy Response Prediction in Early Breast Cancer
Acronym: ADAPT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: West German Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSG-AM06 / ADAPT HR+/HER2-
Record Dates: First submitted 2013-01-25; First posted 2013-01-30 (Estimated); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Cyclophosphamide; Docetaxel; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anthracycline - Taxane (Active Comparator): Study sites can choose between either Epirubicin (90mg/m²) Cyclophosphamide (600mg/m²) q3w OR Epirubicin (90mg/m²) Cyclophosphamide (600mg/m²) q2w for anthracycline treatment and between either 4 x Docetaxel (100mg/m²) q3w OR 12 x Paclitaxel (80mg/m²) q1w for taxane treatment.
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Paclitaxel
- Taxane - Anthracycline (Experimental): Study sites can choose between either Epirubicin (90mg/m²) Cyclophosphamide (600mg/m²) q3w OR Epirubicin (90mg/m²) Cyclophosphamide (600mg/m²) q2w for anthracycline treatment and between either 4 x Docetaxel (100mg/m²) q3w OR 12 x Paclitaxel (80mg/m²) q1w for taxane treatment.
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Paclitaxel

INTERVENTIONS:
Drug: Epirubicin
Drug: Cyclophosphamide
Drug: Docetaxel
Drug: Paclitaxel

SUMMARY:
Trial for the optimization of risk assessment and therapy success prediction in patients with early breast cancer by the use of biomarkers in advance to therapy decision-making to personalize therapies.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, age at diagnosis 18 years and above (consider patients at 70 years and above for ADAPT Elderly)
* Histologically confirmed unilateral primary invasive carcinoma of the breast
* Clinical T1 - T4 (except inflammatory breast cancer)
* All clinical N (cN)
* No clinical evidence for distant metastasis (M0)
* Known HR status and HER2 status (local pathology)
* Tumor block available for central pathology review
* Performance Status ECOG <= 1 or KI >= 80%
* Negative pregnancy test (urine or serum) within 7 days prior to start of induction treatment in premenopausal patients
* Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements
* The patient must be accessible for treatment and follow-up

Additional Inclusion criteria for patients receiving chemotherapy:

* Laboratory requirements for patients receiving neoadjuvant chemotherapy (within 14 days prior to induction treatment):

  * Leucocytes >= 3.5 x 10^9/L
  * Platelets >= 100 x 10^9/L
  * Hemoglobin >= 10 g/dL
  * Total bilirubin <= 1 x ULN
  * ASAT (SGOT) and ALAT (SGPT) <= 2.5 x UNL
  * Creatinine <= 175 µmol/L (2 mg/dl)
* LVEF within normal limits of each institution measured by echocardiography and normal ECG (within 42 days prior to induction treatment)

Exclusion Criteria:

* Known hypersensitivity reaction to the compounds or incorporated substances
* Prior malignancy with a disease-free survival of < 10 years, except curatively treated basalioma of the skin or pTis of the cervix uteri
* Non-operable breast cancer including inflammatory breast cancer
* Previous or concurrent treatment with cytotoxic agents for any reason after consultation with the sponsor
* Concurrent treatment with other experimental drugs. Participation in another interventional clinical trial with or without any investigational not marketed drug within 30 days prior to study entry
* Male breast cancer
* Concurrent pregnancy; patients of childbearing potential must implement a highly effective (less than 1% failure rate) non-hormonal contraceptive measures during the study treatment
* Breast feeding woman
* Sequential breast cancer
* Reasons indicating risk of poor compliance
* Patients not able to consent

Additional Exclusion Criteria for patients receiving chemotherapy:

* Known polyneuropathy ≥ grade 2
* Severe and relevant co-morbidity that would interact with the application of cytotoxic agents or the participation in the study including acute cystitis and ischuria and chronic kidney disease
* Uncompensated cardiac function
* Inadequate organ function including:

  * Leucocytes < 3.5 x 10^9/l
  * Platelets < 100 x 10^9/l
  * Bilirubin above normal limits
  * Alkaline phosphatase >= 5 x UNL
  * ASAT and/or ALAT associated with AP > 2.5 x UNL

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4936 (Estimated)
Dates: Start 2012-05 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Identification of a responder sub-population with intermediate and high risk, which due to therapy has outcome comparable to HR+/RS≤11 | 3 Years

SECONDARY OUTCOMES:
Overall survival | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Harbeck, Prof. Dr., Principal Investigator — Breast Center of the University of Munich (LMU) Universitätsfrauenklinik Großhadern, Munich, Germany; Ulrike Nitz, Prof. Dr., Study Chair — Ev. Krankenhaus Bethesda Brustzentrum Niederrhein, Mönchengladbach, Germany
Locations (2):
- Germany (2):
  - Breast Center of the University of Munich (LMU) Universitätsfrauenklinik Großhadern, Munich, Bavaria
  - Ev. Krankenhaus Bethesda Brustzentrum Niederrhein, Mönchengladbach, North Rhine-Westphalia

REFERENCES:
- [Background] Hofmann D, Nitz U, Gluz O, Kates RE, Schinkoethe T, Staib P, Harbeck N. WSG ADAPT - adjuvant dynamic marker-adjusted personalized therapy trial optimizing risk assessment and therapy response prediction in early breast cancer: study protocol for a prospective, multi-center, controlled, non-blinded, randomized, investigator initiated phase II/III trial. Trials. 2013 Aug 19;14:261. doi: 10.1186/1745-6215-14-261. PMID 23958221
- [Derived] Zhang G, Jurinovic V, Bartels S, Christgen M, Christgen H, Kandt LD, Mishieva L, Ni H, Raap M, Klein J, Katzke AL, Hofmann W, Steinemann D, Kates RE, Gluz O, Graeser M, Kummel S, Nitz U, Plass C, Lehmann U, Zu Eulenburg C, Mansmann U, Gerhauser C, Harbeck N, Kreipe HH. A predictive endocrine resistance index accurately stratifies luminal breast cancer treatment responders and nonresponders. J Clin Invest. 2025 Jul 24;135(19):e177813. doi: 10.1172/JCI177813. eCollection 2025 Oct 1. PMID 40705465
- [Derived] Gluz O, Kuemmel S, Nitz U, Braun M, Ludtke-Heckenkamp K, von Schumann R, Darsow M, Forstbauer H, Potenberg J, Uleer C, Grischke EM, Aktas B, Schumacher C, Zu Eulenburg C, Kates R, Jozwiak K, Graeser M, Wuerstlein R, Baehner R, Christgen M, Kreipe HH, Harbeck N. Nab-paclitaxel weekly versus dose-dense solvent-based paclitaxel followed by dose-dense epirubicin plus cyclophosphamide in high-risk HR+/HER2- early breast cancer: results from the neoadjuvant part of the WSG-ADAPT-HR+/HER2- trial. Ann Oncol. 2023 Jun;34(6):531-542. doi: 10.1016/j.annonc.2023.04.002. Epub 2023 Apr 14. PMID 37062416
- [Derived] Harbeck N, Nitz UA, Christgen M, Kummel S, Braun M, Schumacher C, Potenberg J, Tio J, Aktas B, Forstbauer H, Grischke EM, Scheffen I, Malter W, von Schumann R, Just M, Zu Eulenburg C, Biehl C, Kolberg-Liedtke C, Deurloo R, de Haas S, Jozwiak K, Hauptmann M, Kates R, Graeser M, Wuerstlein R, Kreipe HH, Gluz O; WSG-ADAPT investigators. De-Escalated Neoadjuvant Trastuzumab-Emtansine With or Without Endocrine Therapy Versus Trastuzumab With Endocrine Therapy in HR+/HER2+ Early Breast Cancer: 5-Year Survival in the WSG-ADAPT-TP Trial. J Clin Oncol. 2023 Aug 1;41(22):3796-3804. doi: 10.1200/JCO.22.01816. Epub 2023 Feb 21. PMID 36809046
- [Derived] Nitz UA, Gluz O, Kummel S, Christgen M, Braun M, Aktas B, Ludtke-Heckenkamp K, Forstbauer H, Grischke EM, Schumacher C, Darsow M, Krauss K, Nuding B, Thill M, Potenberg J, Uleer C, Warm M, Fischer HH, Malter W, Hauptmann M, Kates RE, Graser M, Wurstlein R, Shak S, Baehner F, Kreipe HH, Harbeck N. Endocrine Therapy Response and 21-Gene Expression Assay for Therapy Guidance in HR+/HER2- Early Breast Cancer. J Clin Oncol. 2022 Aug 10;40(23):2557-2567. doi: 10.1200/JCO.21.02759. Epub 2022 Apr 11. PMID 35404683
- [Derived] Graeser M, Schrading S, Gluz O, Strobel K, Herzog C, Umutlu L, Frydrychowicz A, Rjosk-Dendorfer D, Wurstlein R, Culemann R, Eulenburg C, Adams J, Nitzsche H, Prange A, Kummel S, Grischke EM, Forstbauer H, Braun M, Potenberg J, von Schumann R, Aktas B, Kolberg-Liedtke C, Harbeck N, Kuhl CK, Nitz U. Magnetic resonance imaging and ultrasound for prediction of residual tumor size in early breast cancer within the ADAPT subtrials. Breast Cancer Res. 2021 Mar 18;23(1):36. doi: 10.1186/s13058-021-01413-y. PMID 33736679
- [Derived] Nitz U, Gluz O, Kreipe HH, Christgen M, Kuemmel S, Baehner FL, Shak S, Aktas B, Braun M, Ludtke-Heckenkamp K, Forstbauer H, Grischke EM, Nuding B, Darsow M, Schumacher C, Krauss K, Malter W, Thill M, Warm M, Wuerstlein R, Kates RE, Harbeck N. The run-in phase of the prospective WSG-ADAPT HR+/HER2- trial demonstrates the feasibility of a study design combining static and dynamic biomarker assessments for individualized therapy in early breast cancer. Ther Adv Med Oncol. 2020 Nov 23;12:1758835920973130. doi: 10.1177/1758835920973130. eCollection 2020. PMID 33281950